CLINICAL TRIAL: NCT02699684
Title: One Month Clinical Comparison of Two Lotrafilcon B Spherical Lenses With Different Packaging Solutions
Brief Title: Comparison of Lotrafilcon B Lenses With Different Packaging Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CLE270-P001
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOHG, then AOA (Other): Lotrafilcon B contact lenses with EOBO-41 worn first, followed by lotrafilcon B contact lenses worn second. Both products worn bilaterally (in both eyes) for 30 days and removed nightly for care using a hydrogen peroxide-based lens care solution.
  Interventions: Device: Lotrafilcon B contact lenses with EOBO-41; Device: Lotrafilcon B contact lenses; Device: Hydrogen peroxide-based lens care solution; Device: Saline solution for rinsing contact lenses; Device: Saline solution for rinsing contact lens case
- AOA, then AOHG (Other): Lotrafilcon B contact lenses worn first, followed by lotrafilcon B contact lenses with EOBO-41 worn second. Both products worn bilaterally for 30 days and removed nightly for care using a hydrogen peroxide-based lens care solution.
  Interventions: Device: Lotrafilcon B contact lenses with EOBO-41; Device: Lotrafilcon B contact lenses; Device: Hydrogen peroxide-based lens care solution; Device: Saline solution for rinsing contact lenses; Device: Saline solution for rinsing contact lens case

INTERVENTIONS:
Device: Lotrafilcon B contact lenses with EOBO-41 — Lotrafilcon B contact lenses packaged with copolymer 845 and EOBO-41
  Other Names: AIR OPTIX® plus HYDRAGLYDE®; AOHG
Device: Lotrafilcon B contact lenses — Lotrafilcon B contact lenses packaged with copolymer 845
  Other Names: AIR OPTIX® AQUA; AOA
Device: Hydrogen peroxide-based lens care solution — Commercially-available hydrogen peroxide-based lens care solution for cleaning, disinfecting, and storing silicone hydrogel soft contact lenses
  Other Names: AOSEPT® PLUS; CLEAR CARE® PLUS
Device: Saline solution for rinsing contact lenses — Commercially-available saline solution used as needed
  Other Names: Minims®
Device: Saline solution for rinsing contact lens case — Commercially-available solution used as needed
  Other Names: LENS PLUS® OCUPURE™

SUMMARY:
The purpose of this study is to evaluate AIR OPTIX® plus HYDRAGLYDE® (AOHG) contact lenses compared to AIR OPTIX® AQUA (AOA) contact lenses in overall lens fit.

DETAILED DESCRIPTION:
Subjects must not wear any contact lenses prior to the visit on Day 1 (Insertion) for Period 1 or Day 1 (Insertion) for Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Must sign Informed Consent Document;
* Manifest cylinder less than or equal to 0.75 Diopter (D) in each eye;
* Successful current wearer (during the past 2 months for a minimum of 5 days per week and 8 hours per day) of AOA contact lenses within the protocol-specified power range;
* Willing to answer text messages on a daily basis during the study;
* Willing to discontinue artificial tears and rewetting drops on the days of study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Habitual lens wear in an extended wear modality (routinely sleeping in lenses overnight for 1 night per week);
* Any anterior segment infection, inflammation, disease or abnormality that contraindicates contact lens wear (within 7 days of enrollment, or current);
* History of herpetic keratitis, corneal surgery or irregular cornea;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Pregnant or lactating;
* Participation in any clinical study within 30 days of Visit 1;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, EMEA, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the United Kingdom (UK).
Pre-assignment Details: Of the 82 enrolled, 6 subjects were exited as screen failures prior to randomization. One subject withdrew consent after randomization, but before exposure to product. This reporting group includes all randomized and exposed subjects (75).
Period: Period 1, First 30 Days of Wear
Arm/Group | AOHG, Then AOA | AOA, Then AOHG
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0
Period: Period 2, Second 30 Days of Wear
Arm/Group | AOHG, Then AOA | AOA, Then AOHG
Started | 37 | 38
Completed | 36 | 38
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and exposed subjects (Full Analysis Set).
Groups:
- Overall: Lotrafilcon B contact lenses with EOBO-41 and lotrafilcon B contact lenses worn bilaterally during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Satisfying the "no Re-fit" Criteria in Both Eyes
Description: Overall lens fit was graded by the Investigator on a 5-point scale: -2 (unacceptably tight); -1 (acceptably tight); 0 (optimal fit); +1 (acceptable loose); +2 (unacceptable loose). 'No re-fit' criteria was satisfied if an acceptable or optimal overall lens fit, that was also within one grade of the habitual lens fit value, was achieved.
Time Frame: Day 30, each product
Population: Full Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Number; unit: percentage of subjects
Groups:
- AOHG Contact Lenses: Lotrafilcon B contact lenses with EOBO-41 worn bilaterally for 30 days in Period 1 or 2, as randomized
- AOA Contact Lenses: Lotrafilcon B contact lenses worn bilaterally for 30 days in Period 1 or 2, as randomized
Arm/Group | AOHG Contact Lenses | AOA Contact Lenses
Number analyzed (Participants) | 75 | 74
percentage of subjects | 93.3 | 94.6

2. Secondary Outcome: Mean Ex Vivo Total Cholesterol Uptake After 30 Days of Wear
Description: The contact lens was removed from the eye. Cholesterol deposits were extracted and measured in micrograms (μg) per lens. Lower deposits indicate increased lens performance. Only one eye (right eye) contributed to the analysis.
Time Frame: Day 30, each product
Population: Full Analysis Set. Only the right (OD) lenses were collected from a subset of subjects.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | AOHG Contact Lenses | AOA Contact Lenses
Number analyzed (Participants) | 32 | 32
μg | 0.44 (0.231) | 0.27 (0.173)

3. Secondary Outcome: Change From Insertion in Minimum Protected Area (MPA)
Description: MPA (the minimum area of the contact lens surface (expressed in %) protected by the tear film between two natural blinks) was assessed by the Investigator during the interblink period using the Tearscope® lighting system. Higher values indicate a more stable tear film in front of the lens. This Outcome Measure was pre-specified for AOHG only. Both eyes contributed to the analysis.
Time Frame: Hour 0 (Lens Insertion) to Hour 12 on Day 1
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: percentage of contact lens surface area
Units Other Than Participants: Eyes
Arm/Group | AOHG Contact Lenses
Number analyzed (Participants) | 45
Number analyzed (Eyes) | 90
percentage of contact lens surface area
  Insertion (Hour 0) | 86.839 (24.775)
  Change from Insertion (Hour 12 - Hour 0) | 4.396 (23.060)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 74 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- AOHG Contact Lenses: All subjects exposed to AOHG contact lenses
- AOA Contact Lenses: All subjects exposed to AOA contact lenses
Arm/Group | Pretreatment | AOHG Contact Lenses | AOA Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/82 | 1/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/82 | 0/75 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=82) | AOHG Contact Lenses (N=75) | AOA Contact Lenses (N=75)
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.